CLINICAL TRIAL: NCT05150678
Title: EXCISION of CAESAREAN SECTION SKIN SCAR AND SUBCUTANEOUS RELEASE VERSUS NON REMOVAL IN REPEATED CAESAREAN SECTION.
Brief Title: Removal Versus Non Removal of Ceserean Section Scar .
Acronym: cs
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, mayada aboelmagd mohamed, principle investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: obstetric and gynacology
Record Dates: First submitted 2021-09-17; First posted 2021-12-09 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2021-11

CONDITIONS: Cesarean Wound; Dehiscence

STUDY DESIGN:
Intervention Model Description: there are two gruops in the study ;one with removal of the scar 2nd with non removal in repeated cs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- removal of cs scar (Experimental): gruop 1 will remove the scar
  Interventions: Procedure: removal of ceserean section scar; Procedure: non removal of cesearean section scar
- non removal of the scar (Experimental): gruop2 will not remove the scar
  Interventions: Procedure: removal of ceserean section scar; Procedure: non removal of cesearean section scar

INTERVENTIONS:
Procedure: removal of ceserean section scar — we will remove the previous scar in group A
Procedure: non removal of cesearean section scar — we will open in the previous cesearean scar in group B

SUMMARY:
EXCISION of cs section skin scar and subcutaneous release versus non removal in repeated cs .aRandomized controlled trial .

DETAILED DESCRIPTION:
All eligible participants will randimized into two groups ; gruop 1 skin removal in which we will going to remove skin scar gruop 2 skin non removal ;direct open in the middle of the previous scar Follow up will be recorded for each participant aphoto will be taken postoperative to score the healing of the wound the follow up will be at one week ,then one month ,then three month acomparison between the two groups will be done .

ELIGIBILITY:
Inclusion Criteria:

1. women with repeated ceserean section
2. pregnant women >32 wk

Exclusion Criteria:

* DM bleeding tendency preeclampsia previous history of wound infection chronic steroid use women refused to participate in Randomized clinical trial

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2022-04 (Estimated); Primary Completion 2023-11 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
the healing score | through the study duration AVERAGE ONE YEAR.
  we will follow up the scar postoperative to compare the healing score by observer scar assessment scale maximaum score 5and patient scar assessment scale.maximum score 10.means WORST scale .

SECONDARY OUTCOMES:
the cosmotic appereance of the scar | through the study duration an average one year
  we will follow up the scar healing postoperative by the observer scale assessment score and the patient scar assessment scale .

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Altman AD, Allen VM, McNeil SA, Dempster J. Pfannenstiel incision closure: a review of current skin closure techniques. J Obstet Gynaecol Can. 2009 Jun;31(6):514-520. doi: 10.1016/S1701-2163(16)34213-X. PMID 19646316
- [Background] Kawakita T, Landy HJ. Surgical site infections after cesarean delivery: epidemiology, prevention and treatment. Matern Health Neonatol Perinatol. 2017 Jul 5;3:12. doi: 10.1186/s40748-017-0051-3. eCollection 2017. PMID 28690864